CLINICAL TRIAL: NCT05347212
Title: Phase II Trial of Immunotherapy in Patients With Carcinomas Arising From the Renal Medulla
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0684; NCI-2022-03632 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Carcinomas; Renal Medullary Carcinoma
MeSH Terms: conditions — Carcinoma | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+Relatlimab (Experimental): nivolumab 480 mg IV plus relatlimab 480 mg IV every 4 weeks for up to 2 years
  Interventions: Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Given by IV
  Other Names: BMS-936558; Opdivo
Drug: Relatlimab — Given by IV
  Other Names: BMS-986016

SUMMARY:
To learn if the combination of nivolumab and relatlimab can help to control renal medullary carcinoma (RMC) that is locally advanced or metastatic (has spread).

DETAILED DESCRIPTION:
OBJECTIVES

Primary objective:

To determine the objective response rate (ORR) of patients with locally advanced or metastatic RMC treated with combination nivolumab plus relatlimab. ORR is defined as the proportion of patients with a best response of complete response (CR) or partial response (PR) by the Response Evaluation Criteria. In Solid Tumors (RECIST 1.1) criteria recorded between Day 1 of the study and the date of objectively documented progression per RECIST 1.1 or the date of subsequent anti-cancer therapy, whichever occurs first. Our goal is to significantly improve the ORR compared with the historical ORR of 29% achieved in our institution using conventional cytotoxic chemotherapies.

Secondary objectives:

* To determine the efficacy and safety of the combination of nivolumab plus relatlimab in patients with RMC. Efficacy will be measured by overall survival (OS), progression-free survival (PFS), time to ORR, duration of response, and the disease control rate (DCR).
* To evaluate potential biomarkers for patient stratification and treatment response, as well as tumor antigen-specific immune responses, such as antibody and T cell responses, as surrogates for anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced or metastatic RMC histologically confirmed by expert pathology review and loss of SMARCB1 staining by immunohistochemistry. Patients with advanced or metastatic unclassified renal cell carcinoma with medullary phenotype (a rare SMARCB1 negative RMC variant occurring in individuals without sickle hemoglobinopathies) are also eligible.
2. Patients will be eligible regardless of whether they have had prior nephrectomy or still have their primary tumor in-situ.
3. Patients must have at least one measurable site of disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures ≥ 15 mm with conventional techniques or ≥ 10 mm with more sensitive techniques such as MRI or CT scan. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
4. Patients should be willing to provide a newly obtained fresh core biopsy of a tumor lesion. Not required if there is a recently obtained fresh specimen on an IRB approved correlated trial up to 6 weeks (42 days) prior to initiation of treatment on Day 1.
5. Patients can be either naïve for any previous systemic treatment or have had any number of prior systemic therapies. However, patients must not have received prior anticancer therapy with antiPD1, anti-PD-L1, anti-CTLA-4, or anti-LAG-3 immune checkpoint inhibitors.
6. There must be evidence of progression on or after last treatment regimen received.
7. ECOG performance status 0-2

   o NOTE: If subject is unable to walk due to paralysis, but is mobile in a wheelchair, subject is considered to be ambulatory for the purpose of assessing their performance status.
8. Age (at the time of consent/assent): ≥ 18 years
9. Consent to MD Anderson companion laboratory protocol 2014-0938
10. Within 14 days of the first dose of the study drugs (cycle 1 day 1), patients must have adequate organ and marrow function as defined below:

    * Hemoglobina ≥9 g/dl (treatment allowed)
    * Absolute neutrophil countb ≥1,000/µL
    * Platelets ≥75,000/µL
    * total bilirubin ≤ 1.5 mg/dl
    * AST(SGOT) or ALT (SGPT) ≤ 2.5 X institutional ULN, except in known hepatic metastasis, wherein may be ≤ 5 x ULN
    * Serum Creatininec ≤ 1.5 x ULN by gender (as long as patient does not require dialysis) aMay receive transfusion b Without growth factor support (filgrastim or pegfilgrastim) for at least 14 days c If creatinine is not <1.5×ULN, then calculate by Cockcroft-Gault methods or local institutional standard and CrCl must be >30 mL/kg/1.73 m2 11 INR and PTT ≤ 1.5 x ULN prior to registration for treatment. Therapeutic anticoagulation with warfarin is allowed if target INR ≤ 3 on a stable dose of warfarin or on a stable dose of low molecular weight (LMW) heparin for > 2 weeks (14 days) at the time of registration for treatment.

      12 Patients with controlled brain metastases are allowed on protocol if they had solitary brain metastases that was surgically resected or treated with radiosurgery or Gamma knife, without recurrence or edema for 1 month (4 weeks). 13 Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of the study drug. 14 Women must not be breastfeeding. 15 WOCBP must agree to follow instructions for method(s) of contraception from the time of registration for treatment for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 30 days (duration of ovulatory cycle) for a total of 5 months post treatment completion. Men must agree to effective contraception from the time of registration for treatment to 7 months post last treatment with nivolumab. 16 WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing as described in these sections.

Exclusion Criteria:

1. Patients must not have any other malignancies within the past 2 years except for in situ carcinoma of any site, or adequately treated (without recurrence post-resection or post-radiotherapy) carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
2. Patients currently receiving anticancer therapies or who have received anticancer therapies (including chemotherapy and targeted therapy) within 2 weeks (14 days) prior to study Day 1 are excluded. Patients who have completed palliative radiation therapy more than 14 days prior to the first dose of the combination immunotherapy are eligible.
3. Patients with persistent grade ≥2 adverse events from prior systemic therapies that would confound timely detection of immune-related adverse events or otherwise hinder patient participation in the clinical trial.
4. Patients, who have had a major surgery or significant traumatic injury (injury requiring > 4 weeks (28 days) to heal) within 4 weeks (28 days) of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that are expected to require major surgery, other than cytoreductive nephrectomy ± retroperitoneal lymph node dissection, during the course of the study.
5. Patients who have organ allografts.
6. Known or suspected autoimmune disease. Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study. Patientswith a history of Hashimoto's thyroiditis only requiring hormone replacement, Type I diabetes, or psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are allowed to participate.
7. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
8. Positive test for hepatitis B virus (HBV) using HBV surface antigen (HBVsAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection. If hepatitis C antibody test is positive then active infection has to be confirmed by hepatitis C RNA testing for the patient to be excluded.
9. Any underlying medical condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea, uncontrolled nausea or vomiting. Patients with active COVID-19 disease as indicated by a positive polymerase reaction (PCR) test are excluded.

   Patients with previous COVID-19 disease are allowed if ≥30 days from last positive test, and COVID-19 symptoms have resolved and/or PCR test is now negative
10. Patients must not have received prior anticancer therapy with anti-LAG-3 immune checkpoint inhibitors.
11. Patients receiving any concomitant systemic therapy for renal cell cancer are excluded.
12. Patients must not be scheduled to receive another experimental drug while on this study.
13. Patients who are on high dose steroid (e.g., > 10mg prednisone daily or equivalent) or other more potent immune suppression medications (e.g., infliximab). Topical, inhaled, intra-articular, ocular, or intranasal corticosteroids (with minimal systemic absorption) are allowed. A brief course (<48 hours) of systemic corticosteroids for prophylaxis (eg, from contrast dye allergy) is permitted.

    Physiological corticosteroid replacement therapy for adrenal insufficiency is also permitted.
14. Troponin T (TnT) or I (TnI) > 2 × institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if a repeat levels within 24 hours are ≤ 1 x ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. Notification of the decision to enroll the participant following cardiologist recommendation has to be made to the MD Anderson Medical Monitor or designee.
15. Left ventricular ejection fraction (LVEF) assessment with documented LVEF < 50% by either transthoracic echocardiogram (TTE) or multigated acquisition (MUGA) scan (TTE preferred test) within 6 months prior to start of study treatment.
16. Active myocarditis, regardless of etiology.
17. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    1. Symptomatic congestive heart failure of New York heart Association Class III or IV
    2. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
    3. Severely impaired lung function as defined as 02 saturation that is 92% or less at rest on room air
    4. Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN (if unfasted glucose elevation, treating physician will evaluate per standard of care)
    5. Systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement) despite appropriate antibiotics or other treatment
    6. Known active or symptomatic viral hepatitis or chronic liver disease. Uncontrolled adrenal insufficiency
    7. Patients with a history of major psychiatric illness judged unable to fully understand the investigational nature of the study and the risks associated with the therapy.
18. Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of nivolumab or relatlimab or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
19. Patients should not receive immunization with attenuated live vaccines within one week (7 days) of registration for treatment or during study period.

    a. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
20. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
21. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods as defined above.
22. Any patients who cannot be compliant with the appointments required in this protocol must not be enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
To establish the objective response rate (ORR) of patients with locally advanced or metastatic RMC treated with combination nivolumab plus relatlimab. | through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Pavlos Msaouel, MD,PHD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org